CLINICAL TRIAL: NCT03615573
Title: Determining the Financial Impact of Breast Cancer Treatment Over a One Year Period for Patients at a Rural Cancer Center
Brief Title: Survey Study: Financial Impact of Breast Cancer Treatment
Status: Completed | Type: Observational
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 1808-42
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quality of Life Surveys — Patients with breast cancer diagnosis complete questionnaires over 20-30 minutes at baseline and at 3, 6, and 12 months after enrollment.

SUMMARY:
A survey study to evaluate the financial impact of breast cancer as self-reported by breast cancer patients over a period of 1 year. The study will also look at the health insurance literacy and patient's utilization of support services.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosed with breast cancer or a recurrence of breast cancer within the past 2 years
* Willing to sign consent
* Able to read and complete surveys in English

Exclusion Criteria:

* Cancer diagnosis other than breast cancer
* More than 2 years since diagnosis with breast cancer or recurrence

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients seen at rural cancer center with diagnosis of breast cancer or a recurrence of breast cancer within the past 2 years
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Change in level of self-reported financial burden | Baseline through 1 year
  Will evaluate the change in Comprehensive Score for Financial Toxicity (COST-FACIT) measurements from baseline to 1 year follow up. This survey consists of 14 questions related to finances.Responses include 5 options with lower scores representing worse outcomes. Scores at 1 year will be compared to baseline scores.

SECONDARY OUTCOMES:
Change in level of self-reported health insurance literacy | Baseline through 1 year
  Will evaluate the change in Health Insurance Literacy Measurements (HILM) from baseline to 1 year follow up
Self-reported access and utilization of institutional support services | Baseline through 1 year
  Will evaluate reported access and utilization of institutional support services and its association to financial burden in the first 12 months after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Perry-Keaty, RN FNP AOCNP, Principal Investigator — The Guthrie Clinic
Locations (1):
- Guthrie Medical Group, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No